CLINICAL TRIAL: NCT01566695
Title: A Phase 3, Multicenter, Randomized, Double-blind Study to Compare the Efficacy and Safety of Oral Azacitidine Plus Best Supportive Care Versus Placebo Plus Best Supportive Care in Subjects With Red Blood Cell Transfusion-dependent Anemia and Thrombocytopenia Due to IPSS Lower-risk Myelodysplastic Syndromes.
Brief Title: The Efficacy and Safety of Oral Azacitidine Plus Best Supportive Care Versus Placebo and Best Supportive Care in Subjects With Red Blood Cell (RBC) Transfusion-Dependent Anemia and Thrombocytopenia Due to International Prognostic Scoring System (IPSS) Low Risk Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AZA-MDS-003; 2012-002471-34 (EudraCT Number)
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Results first posted 2020-02-26 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Azacitidine; cc-486

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral Azacitidine (Experimental): Arm 1: Oral azacitidine tablets 300 mg daily (QD) + best supportive care (BSC) on days 1 through 21 of each 28-day treatment cycle.
  Interventions: Drug: Oral Azacitidine; Other: Best Supportiv Care (BSC)
- Placebo (Placebo Comparator): Arm 2: Identically matching placebo tablets plus best supportive care on days 1 to 21 of each 28-day treatment cycle.
  Interventions: Drug: Placebo; Other: Best Supportiv Care (BSC)

INTERVENTIONS:
Drug: Oral Azacitidine — 300 mg daily, days 1 to 21 of each 28-day treatment cycle
  Other Names: CC-486
  Arms: Oral Azacitidine
Drug: Placebo — Identically matching placebo tablets on day 1 to 21 of each 28-day treatment cycle.
  Arms: Placebo
Other: Best Supportiv Care (BSC) — BSC included and was not limited to packed RBC (packed red blood cell [pRBC] and whole blood), platelet transfusions (single donor or pooled donor), antibiotic, antiviral and/or antifungal therapy, nutritional support, and granulocyte colony stimulating factors (G-CSF) for participants who experienced neutropenic fever/infections.

SUMMARY:
Evaluation of the Efficacy and Safety of Oral Azacitidine plus Best Supportive care versus Placebo and Best Supportive care in subjects with red blood cell (RBC) transfusion-dependent anemia and thrombocytopenia due to International Prognostic Scoring System (IPSS) lower risk myelodysplastic syndromes (MDS).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Have a documented diagnosis of MDS
* Anemia that requires red blood cell transfusions
* Thrombocytopenia (sustained for at least 21 days) within 14 days prior to randomization
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Must agree to follow pregnancy precautions as required by protocol.
* Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures being conducted

Exclusion Criteria:

* Secondary or hypoplastic MDS or other subtype with eligibility for treatment with immunotherapy
* Prior treatment with azacitidine, decitabine, other hypomethylating agents and lenalidomide (for lenalidomide : unless the last dose received is >= 8 weeks prior to inclusion into the study).
* Prior allogeneic or autologous stem cell transplant
* Eligible for allogenic or autologous stem cell transplant
* History of inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis), celiac disease (ie, sprue), prior gastrectomy or upper bowel removal, or any other gastrointestinal disorder or defect
* Thrombocytopenia secondary to other possible causes, including medication(s), congenital disorder(s), immune disorder(s), or microvascular disorder(s)
* Use of cytotoxic, chemotherapeutic, targeted or investigational agents/therapies, thrombopoiesis-stimulating agents (TSAs), erythropoiesis-stimulating agents (ESAs) and other red blood cell hematopoietic growth factors, and within 28 days prior to randomization
* Ongoing medically significant adverse events from previous treatment, regardless of the time period
* Concurrent use of iron-chelating agents, (except for subjects on a stable or decreasing dose for at least 8 weeks (56 days) prior to randomization), corticosteroid (except for subjects on a stable or decreasing dose for ≥ 1 week prior to randomization for medical conditions other than MDS)
* Prior history of cancer, other than MDS, unless the subject has been free of the disease for ≥ 3 years. (Basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, carcinoma in situ of the breast, and incidental histologic finding of prostate cancer) (T1a or T1b using the tumor, nodes, metastasis [TNM] clinical staging system is allowed)
* Significant active cardiac disease within the previous 6 months
* Uncontrolled systemic fungal, bacterial, or viral infection
* Known Human Immunodeficiency Virus (HIV) or Hepatitis C (HCV) infection, or evidence of active Hepatitis B Virus (HBV) infection
* Known clinically significant anemia due to iron, vitamin B12, or folate deficiencies, or autoimmune or hereditary hemolytic anemia, or gastrointestinal bleeding
* Abnormal coagulation parameters
* Abnormal liver function test results
* Abnormal kidney function test results
* Known or suspected hypersensitivity to azacitidine or mannitol
* Any significant medical condition, laboratory abnormality, or psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2013-04-26 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2023-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (196):
- United States (40):
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - Tower Hematology/Oncology Medical Group and Tower Cancer Research Found, Beverly Hills, California
  - City Of Hope, Duarte, California
  - California Cancer Associates for Research and Excellence cCARE, Escondido, California
  - Marin Oncology Associates, Greenbrae, California
  - UCSD-Thornton Hospital, La Jolla, California
  - University of Southern California Norris Cancer Center, Los Angeles, California
  - Local Institution - 942, New Haven, Connecticut
  - University of Florida Health Cancer Center at Orlando Health, Orlando, Florida
  - Phoebe Cancer Center of Phoebe Putney Memorial Hospital, Albany, Georgia
  - Robert H Lurie Comprehensive Cancer Center NW Univ, Chicago, Illinois
  - University Of Illinois At Chicago, Chicago, Illinois
  - University Of Chicago Medical Center, Chicago, Illinois
  - Loyola University Chicago, Maywood, Illinois
  - University Of Kansas Medical Center, Kansas City, Kansas
  - University of Louisville, J.G. Brown Cancer Center, Louisville, Kentucky
  - Hematology And Oncology Specialists, Llc, Metairie, Louisiana
  - Johns Hopkins Medicine, Baltimore, Maryland
  - UMASS Memorial Hospital, Worcester, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Jackson Oncology Associates PLLC, Jackson, Mississippi
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Kansas City VA Medical Center University of Kansas Medical Center, Kansas City, Missouri
  - University Of Nebraska Medical Center, Omaha, Nebraska
  - Weill Cornell Medical College - New York - Presbyterian Hospital, New York, New York
  - Icahn School of Medicine at Mount Sinai Medical Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Eastern Institute of Medical Sciences, Greenville, North Carolina
  - University Hospitals of Cleveland Case Medical Center, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Local Institution - 917, Portland, Oregon
  - Penn Medicine: University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Western Pennsylvania Cancer Institute, Pittsburgh, Pennsylvania
  - Brooke Army Medical Center Francis Street Medical Center, Fort Sam Houston, Texas
  - Local Institution - 900, Houston, Texas
  - Local Institution - 924, Houston, Texas
  - Millennium Physicians - Oncology, Houston, Texas
  - VA Commonwealth University - Massey Cancer Center, Richmond, Virginia
  - Local Institution - 904, Seattle, Washington
  - Waukesha Memorial Hospital, Waukesha, Wisconsin
- Australia (12):
  - Local Institution - 137, Garran, Australian Capital Territory
  - Local Institution - 129, Adelaide, South Australia
  - Local Institution - 134, Clayton, Victoria
  - Local Institution - 132, Frankston, Victoria
  - Local Institution - 131, Camperdown
  - Local Institution - 127, Epping, VIC
  - Local Institution - 133, Fitzroy
  - Local Institution - 135, Kogarah
  - Local Institution - 130, Malvern
  - Local Institution - 126, Milton, Brisbane
  - Local Institution - 138, Waratah
  - Local Institution - 136, Woolloongabba
- Belgium (4):
  - Local Institution - 203, Brasschaat
  - Local Institution - 200, Bruges
  - Local Institution - 202, Charleroi
  - Local Institution - 201, Leuven
- Brazil (5):
  - Local Institution - 154, Fortaleza, Ceará
  - Local Institution - 155, Curitiba, Paraná
  - Local Institution - 152, Porto Alegre, Rio Grande do Sul
  - Local Institution - 153, Rio de Janeiro
  - Local Institution - 151, São Paulo
- Canada (8):
  - Local Institution - 182, Edmonton, Alberta
  - Local Institution - 178, Vancouver, British Columbia
  - Local Institution - 183, Barrie, Ontario
  - Local Institution - 180, Hamilton, Ontario
  - Local Institution - 179, Toronto, Ontario
  - Local Institution - 176, Toronto, Ontario
  - Local Institution - 181, Montreal, Quebec
  - Local Institution - 177, Montreal, Quebec
- Czechia (5):
  - Local Institution - 226, Brno, South Moravian
  - Local Institution - 230, Hradec Králové
  - Local Institution - 229, Olomouc
  - Local Institution - 228, Prague
  - Local Institution - 227, Prague
- Denmark (3):
  - Local Institution - 253, Aarhus
  - Local Institution - 252, Odense C
  - Local Institution - 251, Roskilde
- Finland (2):
  - Local Institution - 276, Helsinki
  - Local Institution - 277, Turku
- France (10):
  - Local Institution - 305, Lille
  - Local Institution - 304, Marseille
  - Local Institution - 301, Nantes
  - Local Institution - 308, Paris
  - Local Institution - 307, Pierre-Bénite
  - Local Institution - 302, Rennes
  - Local Institution - 303, Rouen
  - Local Institution - 306, Strasbourg
  - Local Institution - 300, Toulouse
  - Local Institution - 309, Tours
- Germany (10):
  - Local Institution - 350, Dresden
  - Local Institution - 361, Dresden
  - Local Institution - 355, Düsseldorf
  - Local Institution - 359, Düsseldorf
  - Local Institution - 356, Hamburg
  - Local Institution - 353, Keil
  - Local Institution - 351, Leipzig
  - Local Institution - 352, München
  - Local Institution - 357, Tübingen
  - Local Institution - 360, Ulm
- Greece (6):
  - Local Institution - 853, Heraklion, Irakleio
  - Local Institution - 851, Alexandroupoli
  - Local Institution - 852, Athens
  - Local Institution - 855, Athens
  - Local Institution - 850, Athens
  - Local Institution - 854, Pátrai
- Israel (4):
  - Local Institution - 452, Tel Aviv, Tel Aviv
  - Local Institution - 453, Haifa
  - Local Institution - 451, Petah Tikva
  - Local Institution - 454, Tel Litwinsky
- Italy (22):
  - Local Institution - 482, Alessandria
  - Local Institution - 492, Bari
  - Local Institution - 489, Bologna
  - Local Institution - 494, Cagliari
  - Local Institution - 486, Florence
  - Local Institution - 479, Lecce
  - Local Institution - 498, Milan
  - Local Institution - 488, Milan
  - Local Institution - 497, Novara
  - Local Institution - 480, Palermo
  - Local Institution - 495, Pavia
  - Local Institution - 496, Pisa
  - Local Institution - 485, Reggio Calabria
  - Local Institution - 484, Rionero in Vulture
  - Local Institution - 487, Roma
  - Local Institution - 490, Roma
  - Local Institution - 481, Roma
  - Local Institution - 499, Terni
  - Local Institution - 477, Torino
  - Local Institution - 493, Torrette Di Ancona
  - Local Institution - 478, Udine
  - Local Institution - 476, Venezia - Mestre
- Mexico (4):
  - Local Institution - 830, Huixquilucan de Degollado
  - Local Institution - 828, Monterrey
  - Local Institution - 829, Monterrey
  - Local Institution - 827, Tlalpan
- Netherlands (4):
  - Local Institution - 528, Amsterdam
  - Local Institution - 527, Groningen
  - Local Institution - 526, Nijmegen
  - Local Institution - 529, Rotterdam
- Norway (2):
  - Local Institution - 552, Førde
  - Local Institution - 551, Oslo
- Poland (8):
  - Local Institution - 582, Bydgoszcz
  - Local Institution - 576, Gdansk
  - Local Institution - 579, Krakow
  - Local Institution - 581, Lodz
  - Local Institution - 580, Torun
  - Local Institution - 583, Warsaw
  - Local Institution - 577, Warsaw
  - Local Institution - 578, Wroclaw
- Portugal (5):
  - Local Institution - 604, Beja
  - Local Institution - 600, Coimbra
  - Local Institution - 601, Lisbon
  - Local Institution - 603, Lisbon
  - Local Institution - 602, Porto
- South Korea (5):
  - Local Institution - 704, Busan
  - Local Institution - 703, Daegu
  - Local Institution - 701, Seoul
  - Local Institution - 702, Seoul
  - Local Institution - 700, Seoul
- Spain (12):
  - Local Institution - 626, Badalona (Barcelona)
  - Local Institution - 635, Barcelona
  - Local Institution - 625, Barcelona
  - Local Institution - 636, Granada
  - Local Institution - 629, Madrid
  - Local Institution - 634, Madrid
  - Local Institution - 631, Madrid
  - Local Institution - 632, Málaga
  - Local Institution - 628, Oviedo
  - Local Institution - 630, Salamanca
  - Local Institution - 627, Seville
  - Local Institution - 633, Vitoria-Gasteiz, Álava
- Sweden (3):
  - Local Institution - 653, Gothenburg
  - Local Institution - 652, Lund
  - Local Institution - 651, Stockholm
- Turkey (Türkiye) (6):
  - Local Institution - 401, Adana
  - Local Institution - 405, Antalya
  - Local Institution - 403, Istanbul
  - Local Institution - 400, Istanbul
  - Local Institution - 404, Mersin
  - Local Institution - 402, Trabzon
- United Kingdom (16):
  - Local Institution - 685, Oxford, Oxfordshire
  - Local Institution - 687, Aberdeen
  - Local Institution - 691, Birmingham
  - Local Institution - 686, Bristol
  - Local Institution - 689, Cambridge
  - Local Institution - 678, Cardiff
  - Local Institution - 688, Harrow Middlesex
  - Local Institution - 692, Hull
  - Local Institution - 677, Leicester
  - Local Institution - 683, Liverpool
  - Local Institution - 676, London
  - Local Institution - 684, London
  - Local Institution - 679, Manchester
  - Local Institution - 681, Nottingham
  - Local Institution - 690, Sutton in Ashfield
  - Local Institution - 680, Wolverhampton

REFERENCES:
- [Background] Garcia-Manero G, Almeida A, Giagounidis A, Platzbecker U, Garcia R, Voso MT, Larsen SR, Valcarcel D, Silverman LR, Skikne B, Santini V. Design and rationale of the QUAZAR Lower-Risk MDS (AZA-MDS-003) trial: a randomized phase 3 study of CC-486 (oral azacitidine) plus best supportive care vs placebo plus best supportive care in patients with IPSS lower-risk myelodysplastic syndromes and poor prognosis due to red blood cell transfusion-dependent anemia and thrombocytopenia. BMC Hematol. 2016 May 3;16:12. doi: 10.1186/s12878-016-0049-5. eCollection 2016. PMID 27148452
- [Derived] Garcia-Manero G, Santini V, Almeida A, Platzbecker U, Jonasova A, Silverman LR, Falantes J, Reda G, Buccisano F, Fenaux P, Buckstein R, Diez Campelo M, Larsen S, Valcarcel D, Vyas P, Giai V, Oliva EN, Shortt J, Niederwieser D, Mittelman M, Fianchi L, La Torre I, Zhong J, Laille E, Lopes de Menezes D, Skikne B, Beach CL, Giagounidis A. Phase III, Randomized, Placebo-Controlled Trial of CC-486 (Oral Azacitidine) in Patients With Lower-Risk Myelodysplastic Syndromes. J Clin Oncol. 2021 May 1;39(13):1426-1436. doi: 10.1200/JCO.20.02619. Epub 2021 Mar 25. PMID 33764805
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/home

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized at 101 sites globally. The sites were located in: Europe (76), North America (13), Asia/Pacific (10), and Latin America (2). Results are reported as of the data cut-off date of 25 January 2019.
Pre-assignment Details: Participants were stratified by: average baseline (BL) Red Blood Cell (RBC) transfusion requirement (≤ 4 units versus > 4 units of RBC per 28 days), BL platelet transfusion status (dependent or independent), country of enrollment and Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) (0 to 1 versus 2).
Groups:
- Oral Azacitidine Plus Best Supportive Care: Participants received 300 mg oral azacitidine tablets daily (QD) on days 1 to 21 of each 28-day treatment cycle and best supportive care (BSC) which included and was not limited to packed RBC (packed red blood cell [pRBC] and whole blood), platelet transfusions (single donor or pooled donor), antibiotic, antiviral and/or antifungal therapy, nutritional support, and granulocyte colony stimulating factors (G-CSF) for participants who experienced neutropenic fever/infections.
- Placebo Plus Best Supportive Care: Participants received identically matching placebo tablets QD on days 1 to 21 of each 28-day treatment cycle and BSC which included but was not limited to, pRBC and whole blood, platelet transfusions (single donor or pooled donor), antibiotic, antiviral and/or antifungal therapy, nutritional support, and G-CSF for participants who experienced neutropenic fever/infections.
Period: Overall Study
Arm/Group | Oral Azacitidine Plus Best Supportive Care | Placebo Plus Best Supportive Care
Started | 107 | 109
Completed (Ongoing treatment) | 0 | 0
Not Completed | 107 | 109
Not completed — Lack of Efficacy | 1 | 0
Not completed — Adverse Event | 3 | 0
Not completed — Death | 79 | 86
Not completed — Withdrawal by Subject | 13 | 12
Not completed — Lost to Follow-up | 0 | 3
Not completed — Other reasons | 11 | 8

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all participants who were randomized, regardless of whether they received treatment or not.
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Azacitidine Plus Best Supportive Care | Placebo Plus Best Supportive Care | Total
Number analyzed (Participants) | 107 | 109 | 216
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.0 (9.23) | 73.1 (8.36) | 73.0 (8.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 30 | 58
  Male | 79 | 79 | 158
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 96 | 99 | 195
  Black or African American | 1 | 0 | 1
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islanders | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 0 | 0
  Japanese | 0 | 0 | 0
  Other | 8 | 7 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 9 | 13
  Not Hispanic or Latino | 91 | 93 | 184
  Not Reported | 12 | 7 | 19
Myelodysplastic Syndrome (MDS) World Health Organization (WHO) 2008 Classification [Count of Participants; unit: Participants] — The WHO classification recognizes eight subtypes of MDS that are distinguished by the percentage of myeloblasts, presence or absence of ringed sideroblasts (i.e., erythroid precursors with iron deposits surrounding the nucleus), presence of a monocytosis or a deletion 5q.
  Participants
    RA = Refractory Anemia | 4 | 3 | 7
    RN = Refractory Neutropenia | 0 | 0 | 0
    RT = Refractory Thrombocytopenia | 1 | 0 | 1
    RARS = RA with Ringed Sideroblasts | 3 | 2 | 5
    RCMD = R Cytopenia w/ Multilineage Dysplasia | 80 | 73 | 153
    RAEB-1 RA with Excess Blasts - 1 | 17 | 29 | 46
    RAEB-2 RA with Excess Blasts - 2 | 0 | 0 | 0
    MDS-U (MDS-unclassified) | 2 | 2 | 4
    del (5q) MDS Associated with Isolated del 5q | 0 | 0 | 0
International Prognostic Scoring System (IPSS) [Count of Participants; unit: Participants] — The international prognostic scoring system (IPSS) is a standard for risk assessment in primary myelodysplastic syndromes (MDS) that categorizes prognoses taking into account cytogenetics, cytopenias, blasts and blood counts. The IPSS prognostic subgroups consist of low-, intermediate-1-, intermediate-2-, and high-risk groups. The scale is 0-3.5 at 0.5 increments. Scores of 0=Low; 0.5-1.0=Int-1; 1.5-2.0=Int-2; 2.5-3.5=High risk which corresponds to poorer prognosis.
  Participants
    Low | 0 | 0 | 0
    Intermediate 1 (0.5-1.0) | 106 | 109 | 215
    Intermediate 2 (1.5-2.0) | 1 | 0 | 1
    High | 0 | 0 | 0
Average Red Blood Cell Transfusion Requirement (units per 28 days) [Median (Full Range); unit: units per 28 days] — The average red blood cell (RBC) transfusion units per 28 days is derived using transfusion records before randomization date to randomization date - 84 days (if enrolled under original protocol or protocol amendment 1), or to randomization date - 56 days (if enrolled under protocol 2).
  units per 28 days | 3.33 [1.3 to 10.0] | 3.33 [1.3 to 9.5] | 3.33 [1.3 to 10.0]
Hemoglobin [Mean (Standard Deviation); unit: g/dL] | 8.22 (0.988) | 8.04 (0.960) | 8.13 (0.976)
Platelet Count [Mean (Standard Deviation); unit: 10^9 cells/L] | 27.0 (15.97) | 27.9 (18.11) | 27.5 (17.05)
Platelet Transfusion Status [Count of Participants; unit: Participants] — Participants with thrombocytopenia were defined by 2 platelet counts that were ≤ 75 × 10^9/cells/L with a platelet measurement ≥ 21 days apart. For those who were platelet transfusion-dependent at baseline and did not achieve platelet transfusion independence (TI) ≥ 56 days (8 weeks) during study treatment were considered as non-responders. For participants who were not platelet transfusion-dependent at baseline, development of platelet transfusion dependence, ie, ≥ 2 platelet transfusions in any 56-day (8 week) period during study treatment and were considered worse outcome.
  Participants
    Dependent | 30 | 35 | 65
    Independent | 77 | 74 | 151
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG performance status is used to describe a patient's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability (walking, working, etc.). The scale ranges from 0 to 5: 0 = Fully active, no restrictions; 1 = Restricted activity but ambulatory, able to carry out work of a light nature; 2 = Ambulatory and capable of all self-care but unable to carry out work activities; 3 = Capable to only limited self-care, confined to bed or chair more than 50% of waking hours; 4 = Completely disabled, no self-care, confined to bed or chair; 5 = Dead.
  Participants
    Grade 0-1 | 91 | 94 | 185
    Grade 2 | 16 | 15 | 31
    Grade 3 | 0 | 0 | 0
    Grade 4 | 0 | 0 | 0
    Grade 5 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Red Blood Cell (RBC) Transfusion Independence for ≥ 56 Days
Description: RBC transfusion (tfx) independence was defined as the absence of any RBC transfusion during any consecutive "rolling" 56 days within the treatment period. Participants who did not receive any RBC transfusion during a consecutive rolling 56 days (i.e., day 1 to day 56, day 2 to day 57) were considered as a 56-day RBC transfusion independent responder.
Time Frame: Each participant was assessed for at least 56 days or more; from the date of randomization of study drug up to the data cut-off date of 25 January 2019, approximately 5 months.
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Oral Azacitidine and Best Supportive Care: Participants received 300 mg oral azacitidine tablets daily on days 1 to 21 of each 28-day treatment cycle and BSC included and was not limited to pRBC (packed red blood cell [pRBC] and whole blood), platelet transfusions (single donor or pooled donor), antibiotic, antiviral and/or antifungal therapy, nutritional support, and granulocyte colony stimulating factors (G-CSF) for participants who experienced neutropenic fever/infections.
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 107 | 109
Percentage of Participants | 30.8 [22.1 to 39.6] | 11.9 [5.8 to 18.0]
Statistical Analysis 1: Comparison: Oral Azacitidine and Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority; p = 0.0005, Stratified Mantel-Haenszel Chi-squared — 2 sided; Stratified by average baseline (BL) RBC tfx needs: ≤4 vs >4 units of RBC per 28 days; BL platelet tfx status: dependent or ind. &ECOG PS: 0 to 1 vs 2; Rate Difference = 18.9, 95% CI 2-sided [8.3 to 29.6]

2. Secondary Outcome: Duration of RBC Transfusion Independence Among Participants Who Achieved RBC Transfusion Independence for at Least 56 Days
Description: Duration of RBC transfusion independence was analyzed only for participants who achieved RBC transfusion independence of ≥ 56 days on treatment. Duration of RBC transfusion independence was defined as the time from the date transfusion independence is first observed (day 1 of a ≥ 56 days period without a transfusion) until the date the participants had a subsequently documented RBC transfusion. In the event a participant had more than one ≥56 days rolling periods which met the RBC independence criteria, the duration with the longest rolling period was used in the analysis. Participants who maintained RBC TI through the end of the treatment period were censored at the date of treatment discontinuation, death, or 1 day before the start of the subsequent MDS treatment (if any), whichever occurred first, or the particiapnts latest available assessment date in the database if the treatment was still on-going.
Time Frame: From the date of randomization of study drug up to the data cut-off date of 25 January 2019
Population: Intent to Treat population. Participants who achieved RBC transfusion independence of ≥ 56 days on treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 33 | 13
months | 11.1 [8.2 to 26.0] | 12.0 [2.3 to NA] — Could not be estimated due to the low number of events at the time of the analysis.

3. Secondary Outcome: Time to RBC Transfusion Independence for at Least 56 Days Among Participants Who Achieved RBC Transfusion Independence for at Least 56 Days
Description: Time to RBC transfusion independence of ≥ 56 days was defined as the time between randomization and the date onset of transfusion independence was first observed (ie, Day 1 of 56 without any RBC transfusions).
Time Frame: From the date of randomization of study drug up to the data cut-off date of 25 January 2019; median duration of treatment to oral azacitidine was 5.29 months and 5.36 months for placebo
Population: Responders in the intent to treat population who achieved a 56-day TI response
Measure: Median (Full Range); unit: Months
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 33 | 13
Months | 2.37 [0.0 to 10.9] | 2.04 [0.0 to 14.3]

4. Secondary Outcome: Duration of RBC Transfusion Reduction for Participants Who Achieved RBC Transfusion Reduction of at Least 4 Units of RBCs for at Least 8 Weeks
Description: A participant was considered as a RBC transfusion reduction responder if the participant had at least 4 units reduction in transfusion units over any consecutive 56 days period compared to the baseline transfusion units in 56 days.
Time Frame: From the date of randomization of study drug up to the treatment period; up to the data cut-off date of 25 January 2019; median duration of treatment to oral azacitidine was 5.29 months and 5.36 months for placebo
Population: Intent to Treat population; includes participants who achieved RBC transfusion reduction of at least 4 units for at least 8 weeks.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 45 | 34
months | 10.0 [7.1 to 13.3] | 2.3 [2.0 to 5.0]

5. Secondary Outcome: Percentage of Participants Who Achieved RBC Transfusion Independence for ≥ 84 Days
Description: RBC transfusion independence was defined as the absence of any red blood cell (RBC) transfusion during any consecutive "rolling" 84 days within the treatment period. Participants who did not receive any RBC transfusion during a consecutive rolling 84 days (i.e., day 1 to day 84, day 2 to day 85) were considered as a 84-day RBC transfusion independent responder.
Time Frame: as for outcome 4
Population: The ITT population includes all participants who were randomized, regardless of whether they received treatment or not.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 107 | 109
Percentage of Participants | 28.0 [19.5 to 36.5] | 6.4 [1.8 to 11.0]
Statistical Analysis 1: Comparison: Oral Azacitidine and Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority; p < 0.0001, Stratified Mantel-Haenszel; Chi-squared — 2 sided; [statistical method as in outcome 1, analysis 1]; Rate Difference = 21.6, 95% CI 2-sided [11.9 to 31.3]

6. Secondary Outcome: Duration of RBC Transfusion Independence Among Participants Who Achieved RBC Transfusion Independence for at Least 84 Days
Description: Duration of RBC transfusion independence was analyzed only for participants who achieved RBC transfusion independence of ≥ 84 days on treatment. Duration of RBC transfusion independence was defined as the time from the date transfusion independence is first observed (day 1 of a ≥ 84 days period without a transfusion) until the date the participants had a subsequently documented RBC transfusion. In case a participant had more than one ≥84 days rolling periods which met the RBC independence criteria, the duration with the longest rolling period was used in the analysis.
Time Frame: as for outcome 4
Population: Intent to Treat population. Participants who achieved RBC transfusion independence for at least 84 days on treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 30 | 7
months | 11.1 [8.2 to 26.0] | NA [5.0 to NA] — Could not be estimated due to the low number of events at the time of analysis.
Statistical Analysis 1: Comparison: Oral Azacitidine and Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority; p = 0.4347, Two-Sided Unstratified Log Rank Test

7. Secondary Outcome: Time to RBC Transfusion Independence for at Least 84 Days Among Participants Who Achieved RBC Transfusion Independence for at Least 84 Days
Description: Time to RBC transfusion independence of ≥ 84 days was defined as the time between randomization and the date onset of transfusion independence was first observed (ie, Day 1 of 84 without any RBC transfusions).
Time Frame: as for outcome 4
Population: Participants who achieved a 84-day TI response. Responders in the intent to treat population.
Measure: Median (Full Range); unit: Months
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 30 | 7
Months | 2.64 [0.0 to 9.9] | 4.01 [0.5 to 14.3]

8. Secondary Outcome: Percentage of Participants With an Erythroid Hematological Improvement (HI-E) Response According to 2006 IWG Criteria
Description: Erythroid HI-E improvement was defined as a hemoglobin increase of ≥ 1.5 g/dL; or a reduction in units of RBC transfusions by an absolute number of at least 4 RBC transfusions/8 weeks compared with the pretreatment transfusion number in the previous 8 weeks. Only RBC transfusions given for a hemoglobin of ≤ 9.0 g/dL on treatment were counted in the RBC transfusion response evaluation.
Time Frame: as for outcome 4
Population: The ITT population included all participants who were randomized, regardless of whether they received treatment or not.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 107 | 109
Percentage of Participants
  HI-E Response | 43.0 [33.6 to 52.4] | 32.1 [23.3 to 40.9]
  ≥ 1.5 g/dL Hemoglobin Increase | 23.4 [15.3 to 31.4] | 5.5 [1.2 to 9.8]
  RBC Transfusion Reduction | 42.1 [32.7 to 51.4] | 31.2 [22.5 to 39.9]
Statistical Analysis 1: Comparison: Oral Azacitidine and Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority — HI-E; p = 0.1467, Stratified Mantel-Haenszel. Chi-squared; Stratified by average BL RBC tfx needs: ≤4 units versus >4 units; BL platelet tfx status: dependent or independent and ECOG PS: 0 to 1 vs 2; Rate Difference = 10.9, 95% CI 2-sided [-2.0 to 23.7]
Statistical Analysis 2: Comparison: Oral Azacitidine and Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority — ≥ 1.5 g/dL Hemoglobin Increase; p = 0.0002, Stratified Mantel-Haenszel. Chi-squared; [statistical method as in outcome 8, analysis 1]; Rate Diffrence = 17.9, 95% CI 2-sided [8.8 to 26.9]
Statistical Analysis 3: Comparison: Oral Azacitidine and Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority — RBC Transfusion Reduction; p = 0.1431, Stratified Mantel-Haenszel. Chi-squared; [statistical method as in outcome 8, analysis 1]; Rate Difference = 10.9, 95% CI 2-sided [-1.9 to 23.6]

9. Secondary Outcome: Percentage of Participants With a Hematological Improvement Response in Platelets (HI-P) According to 2006 IWG Criteria
Description: HI-P response was defined according to IWG 2006 criteria (Cheson, 2006) and as: 1. Absolute increase of ≥ 30 X 10^9/L for participants^ starting with > 20 X 10^9/L platelets; 2. Increase from < 20 X 10^9/L to > 20 X 10^9/L and by at least 100%. HI-P must have lasted at least 8 weeks.
Time Frame: as for outcome 4
Population: The ITT population included all participants who were randomized, regardless of whether they received treatment or not.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 107 | 109
Percentage of Participants | 24.3 [16.2 to 32.4] | 7.3 [2.4 to 12.2]
Statistical Analysis 1: Comparison: Oral Azacitidine and Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority; p = 0.0007, Stratified Mantel-Haenszel. Chi-squared; [statistical method as in outcome 8, analysis 1]; Rate Difference = 17.0, 95% CI 2-sided [7.5 to 26.4]

10. Secondary Outcome: Percentage of Participants Who Achieved Platelet Transfusion Independence With a Duration of ≥ 8 Weeks (56 Days)
Description: Platelet transfusion independence was defined as the absence of any platelet transfusion during any consecutive "rolling" 56 days during the treatment period, (ie, Day 1 to 56, Day 2 to 57, Days 3 to 58, etc.). Participants were considered platelet transfusion dependent at baseline if they had received ≥ 2 platelet transfusions during the 56 days immediately preceding randomization and had no consecutive 28-day period during which no platelet transfusions were administered.
Time Frame: as for outcome 4
Population: ITT population; includes participants who were baseline platelet transfusion dependent.
Measure: Number; unit: Percentage Participants
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 30 | 35
Percentage Participants | 16.7 | 14.3

11. Secondary Outcome: Time to Platelet Transfusion Independence
Description: Time to platelet transfusion independence was defined as the time between randomization and the first documented date of onset of transfusion independence (ie, Day 1 of 56 without any platelet transfusions).
Time Frame: as for outcome 4
Population: Intent to Treat population; includes participants who achieved platelet transfusion independence for at least 56 days.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 5 | 5
Months | 9.6 [9.6 to 10.9] | NA [NA to NA] — Median, lower and upper range not calculated due to insufficient number of events.

12. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from randomization to death from any cause and was calculated using randomization date and date of death, or date of last follow-up for censored participants. All subjects were followed until drop out (withdrawal of consent from further data collection or lost to follow-up), death, or study closure. Participants who dropped out or were alive at study closure (or at the time of the interim analysis) had their OS times censored at the time of last contact, as appropriate.
Time Frame: From randomization up to death from any cause; up to a maximum of approximately 10 years on study; median duration of treatment to oral azacitidine was 5.29 months and 5.36 months for placebo
Population: Intent to Treat population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 107 | 109
Months | 17.3 [12.9 to 20.8] | 16.7 [12.8 to 24.0]
Statistical Analysis 1: Comparison: Oral Azacitidine and Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Other; p = 0.6257, Log Rank; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.79 to 1.49]; Cox proportional hazards model with stratifies factors

13. Secondary Outcome: Percentage of Participants With a Hematologic Response According to the 2006 IWG Criteria for MDS
Description: Hematologic response was defined as: • A complete response (CR): <5% myeloblasts, and normal maturation of all cell lines; Peripheral blood (PB) shows: hemoglobin >10 g/dL, neutrophils ≥1.0x10^9/L, platelets ≥100x10^9/dL, blasts (0%) • Partial Response (PR): same as CR bone marrow (BM) shows blasts decreased by ≥ 50% over pre-treatment but still > 5%; Cellularity and morphology not relevant • Marrow CR: BM: ≤ 5% myeloblasts and decrease by ≥ 50% over pre-treatment PB • Stable disease (SD): failure to achieve at least PR, but no evidence of progression for > 8 wks • Failure: death during treatment or disease progression • Disease Progression for those with: - Less than 5% blasts: ≥ 50% increase in blasts to > 5% blasts - 5%-10% blasts:≥ 50% increase to > 10% blasts - 10%-20% blasts:≥ 50% increase to > 20% blasts - 20%-30% blasts ≥ 50% increase to > 30% blasts Any of the following: - ≥ 50% decrease from maximum remission/response in granulocytes or platelets
Time Frame: Response was assessed every 3 cycles; up to the data cut-off date of 25 Jan 2019; median duration of exposure to oral azacitidine was 86.0 days and 119.0 days for placebo
Population: Population includes participants with a CR, PR and mCR who had baseline bone marrow blasts > 5%. ITT population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 107 | 109
Percentage of Participants
  Complete Response (CR) | 7.7 | 0
  Partial Response | 0 | 0
  Marrow CR | 23.1 | 4.2
  Stable Disease (SD) | 2.8 | 30.3
  Disease Progression | 62.6 | 46.8
  Failure due to Death | 0.9 | 0.9

14. Secondary Outcome: Percentage of Participants Who Progressed to Acute Myeloid Leukemia (AML)
Description: Participants with a documented diagnosis of AML arising from previous MDS documented diagnosis.
Time Frame: From randomization of study drug to the end up to final data cut-off date of 25 January 2019; maximum follow-up time was 67.9 months for azacitidine and 64.8 months for placebo group
Population: as for baseline characteristics
Measure: Number; unit: Percentage of Participants
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 107 | 109
Percentage of Participants | 7.5 | 16.5

15. Secondary Outcome: Time to Progression to Acute Myeloid Leukemia (AML) Among Participants Who Progressed to AML
Description: Time to AML progression was defined as the time from the date of randomization until the date the subject has documented progression to AML. For participants who had progression to AML documented in MLL central lab report, the earliest sample collection date with the diagnosis of "s-AML arising from previous MDS" was used as the date to AML progression.
Time Frame: From randomization of study drug to progression of AML; up to a maximum of approximately 10 years on study; median duration of treatment to oral azacitidine was 5.29 months and 5.36 months for placebo
Population: The intent-to-treat (ITT) population who progressed to AML.
Measure: Median (Full Range); unit: Months
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 8 | 18
Months | NA [NA to NA] — The Time to AML was not evaluable due to insufficient number of events. | NA [NA to NA] — The Time to AML was not evaluable due to insufficient number of events.

16. Secondary Outcome: Percentage of Participants With Significant Bleeding Events
Description: Clinically significant bleeding event was defined as: any intracranial or retroperitoneal bleed; bleeding requiring transfusions of > 2 units of blood/blood products; bleeding associated with a decrease in hemoglobin of > 2 g/dL; or bleeding from any site requiring transfusions of > 2 units of blood.
Time Frame: From date of randomization until 28 days after the last dose of IP; up to data cut off date of 25 January 2019; median duration of treatment to oral azacitidine was 5.29 months and 5.36 months for placebo
Population: as for baseline characteristics
Measure: Number; unit: Percentage of Participants
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 107 | 109
Percentage of Participants | 8.4 | 9.2

17. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE)
Description: A TEAE was defined as an adverse event that begins or worsens in intensity of frequency on or after the first dose of study drug through 28 days after last dose of study drug. A serious adverse event (SAE) is any: • Death; • Life-threatening event; • Any inpatient hospitalization or prolongation of existing hospitalization; • Persistent or significant disability or incapacity; • Congenital anomaly or birth defect; • Any other important medical event The investigator determined the relationship of an AE to study drug based on the timing of the AE relative to drug administration and whether or not other drugs, therapeutic interventions, or underlying conditions could provide a sufficient explanation for the event. The severity of an AE was evaluated by the investigator according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) (Version 4.0) where Grade 1 = Mild, Grade 2 = Moderate, Grade 3 = Severe, Grade 4 = Life-threatening and Grade 5 = Death.
Time Frame: From first dose of IP up to 28 days after the last dose of IP or until the last study visit; up to a maximum of approximately 6 months on study
Population: The safety population includes all randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 107 | 109
Participants
  ≥ 1 TEAE | 107 | 108
  ≥ 1 TEAE Related to Study Drug | 102 | 54
  ≥ 1 Serious TEAE | 83 | 69
  ≥ 1 Serious TEAE Related to Study Drug | 38 | 8
  ≥ 1 Grade (GR) 3-4 TEAE | 98 | 81
  ≥ 1 Grade 3-4 TEAE Related to Study Drug | 73 | 20
  ≥ 1 Grade (GR) 3-4 Serious TEAE | 79 | 56
  ≥ 1 GR 3-4 Serious TEAE Related to Study Drug | 38 | 5
  ≥ 1 TEAE Leading to Death | 25 | 14
  ≥ 1 TEAE Related to Study Drug Leading to Death | 9 | 2
  ≥ 1 TEAE Leading to Dose Reduction | 31 | 4
  ≥ 1 TEAE Leading to Dose Interruption | 68 | 40
  ≥ 1 TEAE Leading to Dose Interruption/Reduction | 29 | 2
  ≥ 1 TEAE Leading to Treatment Discontinuation | 34 | 31

18. Secondary Outcome: Mean Change From Baseline in the Physical Well-Being Component of the Functional Assessment of Cancer Therapy-Anemia (FACT-An) Endpoints at Cycle 6
Description: The FACT-An questionnaire is a 47-item, cancer specific questionnaire consisting of a core 27 items measuring 4 general domains physical well being (PWG), social/family (SWB), emotional well being (EWB) and Functional Well-Being (FWB) and an additional 20-item anemia questionnaire that measures fatigue associated items and 7 non-fatigue items. The scales are formatted on 1 to 4 pages for self-administration using a 5-point Likert rating scale (0 = Not at all; 1 = A little bit; 2 = Somewhat; 3 = Quite a Bit and 4 = Very much). Also, general health related quality of life (HRQoL), the FACT-An measures the impact of fatigue and other anemia-related symptoms on patient functioning and is used to assess the effect of treatments in various therapeutic areas, including MDS. The instrument and the fatigue and non-fatigue subscales are scored by summing points from all questions, then converting this sum to a 100 point scale; 0 indicates the poorest QOL and 100 denotes the highest QOL.
Time Frame: Baseline to Cycle 6 Day 1
Population: The Health Related Quality of Life (HR-QoL) evaluable population was defined as participants with a non-missing FACT-An Trial Outcome Index (TOI) score at C1D1 and at least one post-baseline assessment visit.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 42 | 49
Units on a Scale | 0.2 (4.12) | -0.8 (3.91)
Statistical Analysis 1: Comparison: Oral Azacitidine and Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority; p = 0.214, t-test, 2 sided; The p-value was calculated based on a pooled 2-sample, 2-sided t-test for the difference in mean change from baseline between treatment groups

19. Secondary Outcome: Mean Change From Baseline in the Social Well-Being Component of the Functional Assessment of Cancer Therapy-Anemia Instrument at Cycle 6
Description: as for outcome 18
Time Frame: Baseline to Cycle 6 Day 1
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 42 | 49
Units on a Scale | -0.4 (3.96) | -1.1 (4.69)
Statistical Analysis 1: Comparison: Oral Azacitidine and Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority; p = 0.446, t-test, 2 sided; [statistical method as in outcome 18, analysis 1]

20. Secondary Outcome: Mean Change From Baseline in the Emotional Well-Being Component of the Functional Assessment of Cancer Therapy-Anemia Instrument at Cycle 6
Description: as for outcome 18
Time Frame: Baseline to Cycle 6 Day 1
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 42 | 49
Units on a Scale | 1.3 (4.33) | 0.2 (4.35)
Statistical Analysis 1: Comparison: Oral Azacitidine and Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority; p = 0.248, t-test, 2 sided; [statistical method as in outcome 18, analysis 1]

21. Secondary Outcome: Mean Change From Baseline in the Functional Well-Being Component of the FACT-An Instrument at Cycle 6
Description: as for outcome 18
Time Frame: Baseline to Cycle 6 Day 1
Population: The FACT-Anemia evaluable population was defined as all ITT participants with a non-missing FACT-An Trial Outcome Index (TOI) score at C1D1 and at least one post-baseline assessment visit.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 42 | 49
Units on a Scale | 0.5 (3.95) | -1.2 (4.45)
Statistical Analysis 1: Comparison: Oral Azacitidine and Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority; p = 0.058, t-test, 2 sided; [statistical method as in outcome 18, analysis 1]

22. Secondary Outcome: Mean Change From Baseline in the Anemia Subscale Within FACT-An Instrument at Cycle 6
Description: as for outcome 18
Time Frame: Baseline to Cycle 6 Day 1
Population: Health Related Quality of Life (HR-QoL) evaluable population was defined as participants with a non-missing FACT-An Trial Outcome Index (TOI) score at C1D1 and at least one post-baseline assessment visit.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 42 | 49
Units on a Scale | 2.9 (11.81) | -0.6 (10.39)
Statistical Analysis 1: Comparison: Oral Azacitidine and Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority; p = 0.130, t-test, 2 sided; [statistical method as in outcome 18, analysis 1]

23. Secondary Outcome: Mean Change From Baseline in the Fatigue-Related Subscale Within the FACT-An Instrument at Cycle 6
Description: as for outcome 18
Time Frame: Baseline to Cycle 6 Day 1
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 42 | 49
Units on a Scale | 2.1 (8.74) | -0.6 (7.84)
Statistical Analysis 1: Comparison: Oral Azacitidine and Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority; p = 0.123, t-test, 2 sided; [statistical method as in outcome 18, analysis 1]

24. Secondary Outcome: Mean Change From Baseline in the Functional Assessment of Cancer Therapy-Anemia Trial Outcome Index (FACT-An TOI) Summary Scale Within the FACT-An Instrument at Cycle 6
Description: The FACT-G and FACT-An score are summed to form the FACT-An total score. The FACT-An Trial Outcome Index (TOI) consists of the summation of a "summary scale" and includes the Physical Well-being, (PWB; 7 items; score range, 0-28), the Functional Well-being (7 items; score range, 0-28) and the Anemia subscale consisting of 20 items on the same five-point scale, with 13 of them measuring fatigue related symptoms (FS) and seven measuring non-FS. The FACT-An TOI has been demonstrated to be a sensitive indicator of clinical outcomes in a number of diseases including MDS. The Fact-TOI score ranges from 0 to 136. Higher scores on all scales of the Fact-An and subscales on the FACT-TOI reflect better quality of life or fewer symptoms.
Time Frame: Baseline to Cycle 6 Day 1
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 42 | 49
Units on a Scale | 3.7 (17.29) | -2.7 (15.45)
Statistical Analysis 1: Comparison: Oral Azacitidine and Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority; p = 0.069, t-test, 2 sided; [statistical method as in outcome 18, analysis 1]

25. Secondary Outcome: Mean Change From Baseline in the Functional Assessment of Cancer Therapy-Anemia-General (FACT-G) Summary Scale Within the FACT-An Instrument at Cycle 6
Description: The FACT-An is a 47-item, cancer-specific questionnaire consisting of a core 27-item general questionnaire (i.e., the Functional Assessment of Cancer Therapy-General [FACT-G]) The FACT-G measures the 4 domains on a 5-point scale ranging from 0 (not at all) to 4 (very much). The 4 domains are: • Physical Well-being (PWB; 7 items; score range, 0-28), • Social/Family Well-being (SWB; 7 items; score range, 0-28), • Emotional Well-being (EWB; 6 items; score range, 0-24), and • Functional Well-being (7 items; score range, 0-28). The FACT-G is a summation composed of a "summary scale" including the PWB, SWB, EWB and FWB. The FACT-G score range is from 0 to 108. For all summary scales including FACT-G, a higher score indicates better HRQoL or lower level of symptoms.
Time Frame: Baseline to Cycle 6 Day 1
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 42 | 49
Units on a Scale | 1.6 (12.00) | -2.9 (12.11)
Statistical Analysis 1: Comparison: Oral Azacitidine and Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority; p = 0.078, t-test, 2 sided; [statistical method as in outcome 18, analysis 1]

26. Secondary Outcome: Mean Change From Baseline in the Functional Assessment of Cancer Therapy-Anemia-Total Score at Cycle 6
Description: The FACT-G and the anemia subscale (AnS) are summed to form the FACT-An total score and the total score ranges from 0 to 188. The FACT-G measures the 4 domains on a 5-point scale ranging from 0 (not at all) to 4 (very much). The 4 domains are: • Physical Well-being (PWB; 7 items; score range, 0-28), • Social/Family Well-being (SWB; 7 items; score range, 0-28), • Emotional Well-being (EWB; 6 items; score range, 0-24), and • Functional Well-being (7 items; score range, 0-28). The AnS consists of 20 items on the same 5-point scale, with 13 of them measuring fatigue-related symptoms (FS) and 7 measuring non-FS. The AnS and FS scores can range from 0-80 and 0-52, respectively. For all domains and summary subscales, a higher score indicates better HRQoL or lower level of symptoms.
Time Frame: Baseline to Cycle 6 Day 1
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 42 | 49
Units on a Scale | 4.5 (21.88) | -3.5 (20.62)
Statistical Analysis 1: Comparison: Oral Azacitidine and Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority; p = 0.073, t-test, 2 sided; [statistical method as in outcome 18, analysis 1]

27. Secondary Outcome: Percentage of Participants With a Clinically Meaningful Improvment (CMI) From Baseline on the Physical Well-Being Domain Within the FACT-An Instrument at Cycle 6
Description: A clinically meaningful improvement or deterioration was defined by domain specific thresholds of change from baseline. The FACT-An questionnaire is a 47-item, cancer specific questionnaire consisting of a core 27 items measuring 4 general domains physical well being, social/family, emotional well being and Functional Well-Being and an additional 20-item anemia questionnaire that measures fatigue and 7 non-fatigue items. The scales are formatted on 4 pages for self-administration using a 5-point Likert rating scale (0 = Not at all; 1 = A little bit; 2 = Somewhat; 3 = Quite a Bit and 4 = Very much). Also, general HRQoL measures the impact of fatigue and other anemia-related symptoms on patient functioning and is used to assess the effect of treatments in various areas, including MDS. The instrument and the fatigue and non-fatigue subscales are scored by summing points from all questions, then converting this sum to a 100 point scale; 0 = the poorest QOL and 100 = the highest QOL.
Time Frame: Cycle 6 Day 1
Population: as for outcome 22
Measure: Number; unit: Percentage of Participants
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 81 | 95
Percentage of Participants | 17.3 | 13.7
Statistical Analysis 1: Comparison: Oral Azacitidine and Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority; p = 0.560, Cochran-Mantel-Haenszel; The p-value was calculated based on the CMH tests for comparing the odds of experiencing CMI between CC-486 versus placebo; Common Odds Raatio = 0.77, 95% CI 2-sided [0.54 to 1.30]; The common odds ratio and the 95% confidence interval (CI) were calculated using CMH tests, stratified by randomization stratification factors, to compare the odds of experiencing clinically meaningful improvement between CC-486 and placebo

28. Secondary Outcome: Percentage of Participants With a Clinically Meaningful Improvment (CMI) From Baseline on the Social Well-Being Domain Within the FACT-An Instrument at Cycle 6
Description: as for outcome 27
Time Frame: Cycle 6 Day 1
Population: as for outcome 22
Measure: Number; unit: Percentage of Participants
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 81 | 95
Percentage of Participants | 11.1 | 14.7
Statistical Analysis 1: Comparison: Oral Azacitidine and Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority; p = 0.480, Cochran-Mantel-Haenszel; [statistical method as in outcome 27, analysis 1]; Common Odds Raatio = 0.72, 95% CI 2-sided [0.29 to 1.78]; [other analysis details as in outcome 27, analysis 1]

29. Secondary Outcome: Percentage of Participants With a Clinically Meaningful Improvment (CMI) From Baseline on the Emotional Well-Being Domain Within the FACT-An Instrument at Cycle 6
Description: as for outcome 27
Time Frame: Cycle 6 Day 1
Population: as for outcome 22
Measure: Number; unit: Percentage of Participants
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 81 | 95
Percentage of Participants | 23.5 | 15.8
Statistical Analysis 1: Comparison: Oral Azacitidine and Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority; p = 0.197, Cochran-Mantel-Haenszel; [statistical method as in outcome 27, analysis 1]; Common Odds Ratio = 1.67, 95% CI 2-sided [0.76 to 3.65]; [other analysis details as in outcome 27, analysis 1]

30. Secondary Outcome: Percentage of Participants With a Clinically Meaningful Improvment (CMI) From Baseline on the Functional Well-Being Domain Within the FACT-An Instrument at Cycle 6
Description: as for outcome 27
Time Frame: Cycle 6 Day 1
Population: as for outcome 22
Measure: Number; unit: Percentage of Participants
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 81 | 95
Percentage of Participants | 14.8 | 8.4
Statistical Analysis 1: Comparison: Oral Azacitidine and Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority; p = 0.121, Cochran-Mantel-Haenszel; [statistical method as in outcome 27, analysis 1]; Common Odds Ratio = 2.14, 95% CI 2-sided [0.82 to 5.57]; [other analysis details as in outcome 27, analysis 1]

31. Secondary Outcome: Percentage of Participants With a Clinically Meaningful Improvment (CMI) From Baseline on the Anemia Subscale Domain Within the FACT-An Instrument at Cycle 6
Description: as for outcome 27
Time Frame: Cycle 6 Day 1
Population: as for outcome 22
Measure: Number; unit: Percentage of Participants
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 81 | 95
Percentage of Participants | 27.2 | 15.8
Statistical Analysis 1: Comparison: Oral Azacitidine and Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority; p = 0.075, Cochran-Mantel-Haenszel; [statistical method as in outcome 27, analysis 1]; Common Odds Ratio = 2.00, 95% CI 2-sided [0.93 to 4.30]; [other analysis details as in outcome 27, analysis 1]

32. Secondary Outcome: Percentage of Participants With a Clinically Meaningful Improvment (CMI) From Baseline in the Fatigue Related Symptoms Subscale Domain Within the FACT-An Instrument at Cycle 6
Description: as for outcome 27
Time Frame: Cycle 6 Day 1
Population: as for outcome 22
Measure: Number; unit: Percentage of Participants
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 81 | 95
Percentage of Participants | 27.2 | 18.9
Statistical Analysis 1: Comparison: Oral Azacitidine and Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority; p = 0.222, Cochran-Mantel-Haenszel; [statistical method as in outcome 27, analysis 1]; Common Odds Ratio = 1.58, 95% CI 2-sided [0.76 to 3.29]; [other analysis details as in outcome 27, analysis 1]

33. Secondary Outcome: Percentage of Participants With a Clinically Meaningful Improvment (CMI) From Baseline in the Functional Assessment of Cancer Therapy-Anemia Trial Outcome Index Subscale Domain Within the FACT-An Instrument at Cycle 6
Description: as for outcome 27
Time Frame: Cycle 6 Day 1
Population: as for outcome 22
Measure: Number; unit: Percentage of Participants
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 81 | 95
Percentage of Participants | 19.8 | 12.6
Statistical Analysis 1: Comparison: Oral Azacitidine and Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority; p = 0.249, Cochran-Mantel-Haenszel; [statistical method as in outcome 27, analysis 1]; Common Odds Ratio = 1.65, 95% CI 2-sided [0.71 to 3.83]; [other analysis details as in outcome 27, analysis 1]

34. Secondary Outcome: Percentage of Participants With a Clinically Meaningful Improvment (CMI) From Baseline in the Functional Assessment of Cancer Therapy-Anemia-General Subscale Domain Within the FACT-An Instrument at Cycle 6
Description: as for outcome 27
Time Frame: Cycle 6 Day 1
Population: The HRQoL evaluable population was defined as participants with a non-missing FACT-An Trial Outcome Index (TOI) score baseline visit and at least one post-baseline assessment visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 81 | 95
Percentage of Participants | 23.5 | 13.7
Statistical Analysis 1: Comparison: Oral Azacitidine and Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority; p = 0.082, Cochran-Mantel-Haenszel; [statistical method as in outcome 27, analysis 1]; Common Odds Ratio = 2.03, 95% CI 2-sided [0.92 to 4.48]; [other analysis details as in outcome 27, analysis 1]

35. Secondary Outcome: Percentage of Participants With a Clinically Meaningful Improvement (CMI) From Baseline in the Functional Assessment of Cancer Therapy Anemia-Total Score Domain Within the FACT-An Instrument at Cycle 6
Description: as for outcome 27
Time Frame: Cycle 6 Day 1
Population: as for outcome 22
Measure: Number; unit: Percentage of Participants
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 81 | 95
Percentage of Participants | 19.8 | 11.6
Statistical Analysis 1: Comparison: Oral Azacitidine and Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority; p = 0.153, Cochran-Mantel-Haenszel; [statistical method as in outcome 27, analysis 1]; Common Odds Ratio = 1.86, 95% CI 2-sided [0.79 to 4.34]; [other analysis details as in outcome 27, analysis 1]

36. Secondary Outcome: Percentage of Participants With Change From Baseline in Responses to the Fact-Anemia Item GP-5 - Cycle 2 Day 1 (C2D1)
Description: The distribution (frequency and percentage) of the observed responses (i.e., "Not at all (0)," "A little bit (1)," "Somewhat (2)," "Quite a bit (3)," "Very much (4)," and missing) to Item GP-5 ("I am bothered by side effects of treatment" in the past seven days) of the FACT-An at each scheduled visit were summarized for each treatment group. The denominator for the percentage calculation per treatment group was based on the number of the FACT-An evaluable population at baseline. The distribution of change in responses (improved [i.e., change score from 1 to 4], no change [0], worsened by one level [-1], worsened by ≥2 levels [-2 to -4], and missing) from baseline at each post-baseline scheduled visit were summarized by treatment group.
Time Frame: From Baseline to Cycle 2 Day 1 (C2D1)
Population: as for outcome 34
Measure: Number; unit: Percentage of Participants
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 81 | 95
Percentage of Participants
  Improved | 2.5 | 10.5
  No Change | 30.9 | 49.5
  Worsened by 1 Level | 25.9 | 23.2
  Worsened by 2 Levels | 23.5 | 6.3
  Missing | 17.3 | 10.5
Statistical Analysis 1: Comparison: Oral Azacitidine and Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority; p < 0.001, Fisher Exact

37. Secondary Outcome: Percentage of Participants With Change From Baseline in Responses to the Fact-Anemia Item GP-5 - Cycle 3 Day 1 (C3D1)
Description: as for outcome 36
Time Frame: From Baseline to Cycle 3 Day 1 (C3D1)
Population: as for outcome 34
Measure: Number; unit: Percentage of Participants
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 81 | 95
Percentage of Participants
  Improved | 7.4 | 10.5
  No Change | 24.7 | 41.1
  Worsened by 1 Level | 16.0 | 18.9
  Worsened by 2 Levels | 23.5 | 13.7
  Missing | 28.4 | 15.8
Statistical Analysis 1: Comparison: Oral Azacitidine and Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority; p = 0.046, Fisher Exact

38. Secondary Outcome: Percentage of Participants With Change From Baseline in Responses to the Fact-Anemia Item GP-5 - Cycle 4 Day 1 (C4D1)
Description: as for outcome 36
Time Frame: From Baseline to Cycle 4 Day 1 (C4D1)
Population: as for outcome 34
Measure: Number; unit: Percentage of Participants
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 81 | 95
Percentage of Participants
  Improved | 2.5 | 9.5
  No Change | 32.1 | 37.9
  Worsened by 1 Level | 16.0 | 14.7
  Worsened by 2 Levels | 14.8 | 6.3
  Missing | 34.6 | 31.6
Statistical Analysis 1: Comparison: Oral Azacitidine and Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority; p = 0.134, Fisher Exact

39. Secondary Outcome: Percentage of Participants With Change From Baseline in Responses to the Fact-Anemia Item GP-5 - Cycle 5 Day 1 (C5D1)
Description: as for outcome 36
Time Frame: From Baseline to Cycle 5 Day 1 (C5D1)
Population: as for outcome 34
Measure: Number; unit: Percentage of Participants
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 81 | 95
Percentage of Participants
  Improved | 2.5 | 7.4
  No Change | 25.9 | 34.7
  Worsened by 1 Level | 13.6 | 12.6
  Worsened by 2 Levels | 8.6 | 5.3
  Missing | 49.4 | 40.0
Statistical Analysis 1: Comparison: Oral Azacitidine and Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority; p = 0.324, Fisher Exact

40. Secondary Outcome: Percentage of Participants With Change From Baseline in Responses to the Fact-Anemia Item GP-5 - Cycle 6 Day 1 (C6 D1)
Description: as for outcome 36
Time Frame: From Baseline to Cycle 6 Day 1 (C6 D1)
Population: as for outcome 34
Measure: Number; unit: Percentage of Participants
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 81 | 95
Percentage of Participants
  Improved | 1.2 | 4.2
  No Change | 25.9 | 27.4
  Worsened by 1 Level | 9.9 | 12.6
  Worsened by 2 Levels | 14.8 | 7.4
  Missing | 48.1 | 48.4
Statistical Analysis 1: Comparison: Oral Azacitidine and Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority; p = 0.442, Fisher Exact

41. Secondary Outcome: Percentage of Participants With Change From Baseline in Responses to the Fact-Anemia Item GP-5 - Cycle 7 Day 1 (C7D1)
Description: as for outcome 36
Time Frame: From Baseline to Cycle 7 Day 1 (C7D1)
Population: as for outcome 34
Measure: Number; unit: Percentage of Participants
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 81 | 95
Percentage of Participants
  Improved | 1.2 | 1.1
  No Change | 25.9 | 21.1
  Worsened by 1 Level | 11.1 | 3.2
  Worsened by 2 Levels | 7.4 | 3.2
  Missing | 54.3 | 71.6
Statistical Analysis 1: Comparison: Oral Azacitidine and Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority; p = 0.063, Fisher Exact

42. Secondary Outcome: Percentage of Participants With Change From Baseline in Responses to the Fact-Anemia Item GP-5 - End of Treatment
Description: as for outcome 36
Time Frame: From Baseline to End of Treatment
Population: as for outcome 34
Measure: Number; unit: Percentage of Participants
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 81 | 95
Percentage of Participants
  Improved | 2.5 | 6.3
  No Change | 14.8 | 25.3
  Worsened by 1 Level | 9.9 | 8.4
  Worsened by 2 Levels | 9.9 | 12.6
  Missing | 63.0 | 47.4
Statistical Analysis 1: Comparison: Oral Azacitidine and Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority; p = 0.198, Fisher Exact

43. Secondary Outcome: Percentage of Participants With Improved, Worsened, or No Change in the European Quality of Life-Five Dimension-Three Level (EQ-5D-3L) Mobility Dimension Responses at Cycle 6
Description: The EQ-5D-3L is a generic, self-administered questionnaire that consists of 5 dimensions: mobility, self-care, pain, usual activities, and anxiety/depression. Each dimension has 3 levels of severity corresponding to no problems, some problems, and extreme problems. It also includes a Visual Analog Scale that recorded the respondent's self-rated health on a vertical, 0-100 scale, where 100 = Best imaginable health state and 0 = Worst imaginable health state. Distribution of the observed responses (i.e., no problems, moderate problems, severe problems, and missing) of the 5 dimensions at each visit was summarized per arm. The denominator for the percentage calculation per group was based on the number of the EQ-5D-3L evaluable population at baseline. The distribution of change in responses (i.e., improved [by ≥1 level], no change, worsened [by ≥1 level], and missing) from baseline are reported.
Time Frame: From Baseline to Cycle 6 Day 1
Population: The HRQoL evaluable population was defined as participants with a EQ-5D-3L health utility at baseline and at least one post-baseline assessment visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 81 | 95
Percentage of Participants
  Improved | 8.6 | 8.4
  No Change | 35.8 | 33.7
  Worsened | 7.4 | 9.5
  Missing | 48.1 | 48.4
Statistical Analysis 1: Comparison: Oral Azacitidine and Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority; p = 0.972, Fisher Exact

44. Secondary Outcome: Percentage of Participants With Improved, Worsened, or No Change in the European Quality of Life-Five Dimension-Three Level of Self-Care Dimension Responses at Cycle 6
Description: as for outcome 43
Time Frame: From Baseline to Cycle 6 Day 1
Population: as for outcome 43
Measure: Number; unit: Percentage of Participants
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 81 | 95
Percentage of Participants
  Improved | 2.5 | 4.2
  No Change | 42.0 | 44.2
  Worsened | 7.4 | 3.2
  Missing | 48.1 | 48.4
Statistical Analysis 1: Comparison: Oral Azacitidine and Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority; p = 0.601, Fisher Exact

45. Secondary Outcome: Percentage of Participants With Improved, Worsened, or No Change in the European Quality of Life-Five Dimension-Three Level Usual Activities Dimension Responses at Cycle 6
Description: TThe EQ-5D-3L is a generic, self-administered questionnaire that consists of 5 dimensions: mobility, self-care, pain, usual activities, and anxiety/depression. Each dimension has 3 levels of severity corresponding to no problems, some problems, and extreme problems. It also includes a Visual Analog Scale that recorded the respondent's self-rated health on a vertical, 0-100 scale, where 100 = Best imaginable health state and 0 = Worst imaginable health state. Distribution of the observed responses (i.e., no problems, moderate problems, severe problems, and missing) of the 5 dimensions at each visit was summarized per arm. The denominator for the percentage calculation per group was based on the number of the EQ-5D-3L evaluable population at baseline. The distribution of change in responses (i.e., improved [by ≥1 level], no change, worsened [by ≥1 level], and missing) from baseline are reported.
Time Frame: From Baseline to Cycle 6 Day 1
Population: as for outcome 43
Measure: Number; unit: Percentage of Participants
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 81 | 95
Percentage of Participants
  Improved | 11.1 | 3.2
  No Change | 28.4 | 41.1
  Worsened | 12.3 | 7.4
  Missing | 48.1 | 48.4
Statistical Analysis 1: Comparison: Oral Azacitidine and Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority; p = 0.070, Fisher Exact

46. Secondary Outcome: Percentage of Participants With Improved, Worsened, or No Change in the European Quality of Life-Five Dimension-Three Level in the Pain/Discomfort Dimension Responses at Cycle 6
Description: as for outcome 43
Time Frame: From Baseline to Cycle 6 Day 1
Population: as for outcome 43
Measure: Number; unit: Percentage of Participants
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 81 | 95
Percentage of Participants
  Improved | 13.6 | 8.4
  No Change | 33.3 | 32.6
  Worsened | 4.9 | 10.5
  Missing | 48.1 | 48.4
Statistical Analysis 1: Comparison: Oral Azacitidine and Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority; p = 0.436, Fisher Exact

47. Secondary Outcome: Percentage of Participants With Improved, Worsened, or No Change in the European Quality of Life-Five Dimension-Three Level in the Anxiety/Depression Dimension Responses at Cycle 6
Description: as for outcome 43
Time Frame: From Baseline to Cycle 6 Day 1
Population: as for outcome 43
Measure: Number; unit: Percentage of Participants
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 81 | 95
Percentage of Participants
  Improved | 4.9 | 7.4
  No Change | 35.8 | 37.9
  Worsened | 11.1 | 6.3
  Missing | 48.1 | 48.4
Statistical Analysis 1: Comparison: Oral Azacitidine and Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority; p = 0.683, Fisher Exact

48. Secondary Outcome: Healthcare Resource Utilization (HRU): Number of Participants Who Were Hospitalized
Description: The number of reasons for hospitalizations and hospital admissions during the treatment period were monitored and include those associated with: AEs, protocol-driven procedures, transfusions, non-protocol procedures, elective procedures or those associated with social, practical or technical reasons in the absence of AEs. HRU was defined as any consumption of healthcare resources directly or indirectly related to the treatment of the patient.
Time Frame: From date of randomization up to 28 days after the last dose of study drug; up to data cut off date of 25 January 2019; median duration of treatment to oral azacitaidine was 5.29 months and 5.36 months for placebo
Population: The safety population includes all randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 107 | 109
Participants
  Adverse Events | 79 | 65
  Protocol Driven Procedures | 2 | 7
  Non-Protocol Driven Procedures | 9 | 19
  Transfusion | 32 | 33
  Procedure Planned Prior to Signing Consent | 0 | 4
  Elective Procedures | 4 | 10
  Social, Technical or Practical Reason except AEs | 4 | 6

49. Secondary Outcome: Healthcare Resource Utilization (HRU): Total Number of Days Hospitalized Due to Any Reason
Description: The total number of days hospitalized due to any reason during the treatment period was monitored. HRU was defined as any consumption of healthcare resources directly or indirectly related to the treatment of the patient.
Time Frame: as for outcome 48
Population: The safety population includes all randomized participants who received at least one dose of study drug.
Measure: Number; unit: Days
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 107 | 109
Days | 3513 | 2688

50. Secondary Outcome: Healthcare Resource Utilization (HRU): Total Number of Days Hospitalized Per Total Patient-Years
Description: The number of days hospitalized per total patient years. HRU was defined as any consumption of healthcare resources directly or indirectly related to the treatment of the patient.
Time Frame: as for outcome 48
Population: The safety population includes all randomized participants who received at least one dose of study drug.
Measure: Number; unit: Days Per Total Patient Years
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 107 | 109
Days Per Total Patient Years | 41.44 | 40.53

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their randomization to study completion, (up to approximately 10 years). SAEs and Other AEs were assessed from first dose to 28 days following last dose (up to approximately 6 months)
Description: Median duration of treatment to oral azacitaidine was 5.29 months and 5.36 months for placebo
Arm/Group | Oral Azacitidine and Best Supportive Care | Placebo Plus Best Supportive Care
All-Cause Mortality (participants affected / at risk) | 83/107 | 86/109
Serious Adverse Events (participants affected / at risk) | 83/107 | 69/109
Other Adverse Events (participants affected / at risk) | 107/107 | 104/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Azacitidine and Best Supportive Care (N=107) | Placebo Plus Best Supportive Care (N=109)
Anaemia (Blood and lymphatic system disorders) | 7 | 5
Blood loss anaemia (Blood and lymphatic system disorders) | 1 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 29 | 9
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 2
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 2 | 2
Cardiac failure congestive (Cardiac disorders) | 3 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 0
Long QT syndrome (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Tachyarrhythmia (Cardiac disorders) | 2 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 2 | 0
Neutropenic colitis (Gastrointestinal disorders) | 1 | 0
Oesophageal achalasia (Gastrointestinal disorders) | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Oral mucosal blistering (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Gait disturbance (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 3 | 1
Hypothermia (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 2 | 0
Pyrexia (General disorders) | 8 | 4
Sudden death (General disorders) | 0 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Arteriovenous fistula site infection (Infections and infestations) | 1 | 0
Atypical pneumonia (Infections and infestations) | 2 | 0
Bacteraemia (Infections and infestations) | 0 | 2
Bronchitis (Infections and infestations) | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 2 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Coronavirus infection (Infections and infestations) | 1 | 0
Cystitis escherichia (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Epididymitis (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0
Febrile infection (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis clostridial (Infections and infestations) | 0 | 1
Groin abscess (Infections and infestations) | 1 | 0
Haemophilus infection (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Klebsiella infection (Infections and infestations) | 1 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 4
Lymph gland infection (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 1 | 0
Meningitis bacterial (Infections and infestations) | 1 | 0
Myringitis (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 5 | 1
Pharyngeal abscess (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 13 | 12
Pneumonia aspiration (Infections and infestations) | 1 | 0
Pneumonia fungal (Infections and infestations) | 2 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Prostatic abscess (Infections and infestations) | 0 | 1
Pseudomonal sepsis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1
Respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 8 | 3
Septic shock (Infections and infestations) | 6 | 3
Skin infection (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 1
Urinary tract infection (Infections and infestations) | 2 | 1
Urinary tract infection bacterial (Infections and infestations) | 1 | 1
Viral sepsis (Infections and infestations) | 1 | 0
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Cystitis radiation (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 4 | 0
Febrile nonhaemolytic transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood urea increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Polychondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carcinoma in situ of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Central nervous system leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mantle cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Myelodysplastic syndrome with excess blasts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transformation to acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 6
Central nervous system lesion (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 2 | 0
IIIrd nerve paresis (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Status epilepticus (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Bipolar disorder (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 2
Acute kidney injury (Renal and urinary disorders) | 2 | 3
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0
Prerenal failure (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 2 | 0
Urinary retention (Renal and urinary disorders) | 1 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Arteritis (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Polyarteritis nodosa (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Azacitidine and Best Supportive Care (N=107) | Placebo Plus Best Supportive Care (N=109)
Anaemia (Blood and lymphatic system disorders) | 23 | 17
Leukopenia (Blood and lymphatic system disorders) | 10 | 3
Neutropenia (Blood and lymphatic system disorders) | 52 | 16
Thrombocytopenia (Blood and lymphatic system disorders) | 30 | 18
Atrial fibrillation (Cardiac disorders) | 7 | 2
Cardiac failure (Cardiac disorders) | 6 | 1
Abdominal pain (Gastrointestinal disorders) | 16 | 14
Constipation (Gastrointestinal disorders) | 51 | 24
Diarrhoea (Gastrointestinal disorders) | 73 | 26
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 1
Gingival bleeding (Gastrointestinal disorders) | 7 | 4
Haemorrhoids (Gastrointestinal disorders) | 4 | 6
Mouth haemorrhage (Gastrointestinal disorders) | 10 | 7
Nausea (Gastrointestinal disorders) | 81 | 25
Rectal haemorrhage (Gastrointestinal disorders) | 3 | 8
Vomiting (Gastrointestinal disorders) | 67 | 11
Asthenia (General disorders) | 25 | 20
Fatigue (General disorders) | 25 | 22
Oedema peripheral (General disorders) | 30 | 17
Pyrexia (General disorders) | 32 | 15
Cellulitis (Infections and infestations) | 6 | 3
Oral herpes (Infections and infestations) | 6 | 3
Pneumonia (Infections and infestations) | 10 | 4
Upper respiratory tract infection (Infections and infestations) | 7 | 4
Urinary tract infection (Infections and infestations) | 12 | 5
Contusion (Injury, poisoning and procedural complications) | 16 | 3
Fall (Injury, poisoning and procedural complications) | 6 | 1
Alanine aminotransferase increased (Investigations) | 10 | 6
Serum ferritin increased (Investigations) | 6 | 5
Weight decreased (Investigations) | 11 | 3
Decreased appetite (Metabolism and nutrition disorders) | 27 | 10
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 6 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 10
Hypomagnesaemia (Metabolism and nutrition disorders) | 11 | 5
Iron overload (Metabolism and nutrition disorders) | 7 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 4
Dizziness (Nervous system disorders) | 8 | 9
Syncope (Nervous system disorders) | 6 | 1
Anxiety (Psychiatric disorders) | 9 | 4
Confusional state (Psychiatric disorders) | 6 | 1
Depression (Psychiatric disorders) | 7 | 2
Insomnia (Psychiatric disorders) | 11 | 6
Haematuria (Renal and urinary disorders) | 4 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 15
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 15
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 28 | 21
Ecchymosis (Skin and subcutaneous tissue disorders) | 6 | 10
Petechiae (Skin and subcutaneous tissue disorders) | 21 | 20
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 8
Haematoma (Vascular disorders) | 11 | 11
Hypertension (Vascular disorders) | 5 | 7
Hypotension (Vascular disorders) | 6 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is > 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 additional days. Investigator must delete confidential information before submission and defer publication to permit patent applications.

DOCUMENTS (2):
  • Study Protocol (2022-05-24): https://cdn.clinicaltrials.gov/large-docs/95/NCT01566695/Prot_002.pdf
  • Statistical Analysis Plan (2019-03-27): https://cdn.clinicaltrials.gov/large-docs/95/NCT01566695/SAP_000.pdf